CLINICAL TRIAL: NCT05295277
Title: Validation of Optical Genome Mapping for the Identification of Constitutional Genomic Variants in a Postnatal Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bionano Genomics (Industry)
Collaborators: University of Rochester (Other); Columbia University (Other); Greenwood Genetic Center (Other); Praxis Genomics (Unknown); Augusta University (Other); Medical College of Wisconsin (Other); University of Iowa (Other)
Responsible Party: Sponsor
Other Study IDs: 20203726
Record Dates: First submitted 2022-03-07; First posted 2022-03-25 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Developmental Disability; Intellectual Disability; Autism Spectrum Disorder; Congenital Anomaly; Fragile X Syndrome; Facioscapulohumeral Muscular Dystrophy 1
Keywords: Validation study; Comparison study; New technology compared to standard of care
MeSH Terms: conditions — Developmental Disabilities; Intellectual Disability; Autism Spectrum Disorder; Congenital Abnormalities; Fragile X Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood or banked lymphoblastoid cell lines (LCLs) will be sent to Bionano Genomics for sample blinding. Specimens are aliquoted, banked, and stored frozen. The specimens will be used for OGM testing or follow up testing using standard of care test methods, as needed and determined by the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of care genetic testing group: Individuals with genomic test results from a standard of care (SOC) test (such as CMA, karyotyping, Southern blot analysis, PCR, FISH, and/or NGS, etc.) will be enrolled in the study to compare the SOC result to results from optical genome mapping.
  Interventions: Other: Standard of care genetic testing group

INTERVENTIONS:
Other: Standard of care genetic testing group — N/A - no intervention as this is an observational study.

SUMMARY:
The purpose of this research use only (RUO) study is to detect genomic structural variants (SVs) in human DNA by Optical Genome Mapping (OGM) using the Bionano Genomics Saphyr system. SVs are a type of genetic alternation that includes deletions, duplications, and both balanced and unbalanced rearrangements (ex: inversions or translocations), as well as specific repeat expansions and contractions. The results of OGM analysis will be compared to prior clinical genetic test results to determine how OGM compares to current standard of care (SOC) clinical test methods such as chromosomal microarray analysis (CMA), karyotyping, Southern blot analysis, polymerase chain reaction (PCR), fluorescence in situ hybridization (FISH), and/or next generation sequencing (NGS), etc.

DETAILED DESCRIPTION:
Optical genome mapping (OGM) is an emerging next-generation cytogenomic tool that enables a comprehensive analysis of structural variants (SVs) in the genome. OGM, in its current iteration, is performed on the Saphyr system, which is developed and marketed by Bionano Genomics (San Diego, CA). OGM employs imaging of ultra-long DNA molecules (>150 kbp) that are labeled at a unique 6 base-pair sequence motif (CTTAAG) that occurs throughout the genome. The images of the labeled DNA molecules are used to generate a de novo assembly that can be compared to a reference genome to identify all classes of SVs, such as deletions, duplications, balanced/ unbalanced genomic rearrangements (insertions, inversions, and translocations), and repeat array expansions/contractions). In addition, a separate coverage-based algorithm enables the detection of genome-wide copy number analysis (similar to CMA), and the absence of heterozygosity (AOH) analysis. In the same assay, a concurrent or stepwise data analysis pipeline allows for sizing pathogenic CGG repeat expansions (consistent with fragile X syndrome) as well as D4Z4 repeat contractions which are consistent with facioscapulohumeral muscular dystrophy type 1 (FSHD1). Recently, in several studies, OGM has demonstrated excellent concordance with standard-of-care testing. Importantly, the OGM workflow can provide results within three-five days.

The aim of this double-blinded, multi-site, retrospective, observational, Institutional Review Board (IRB)-approved study is to evaluate the concordance of structural variant detection by OGM compared to standard of care tests (such as CMA, karyotyping, Southern blot analysis, PCR, FISH, and/or NGS, etc.), in a large cohort containing a variety of SVs including aneuploidies, intragenic and contiguous deletions, duplications, balanced and unbalanced translocations, inversions, isochromosomes, ring chromosomes, repeat expansions, repeat contractions, and more. This study is also designed to assess the sensitivity, specificity, and reproducibility of OGM analysis conducted at multiple sites, by numerous operators, and on different Saphyr instruments. Consensus testing and interpretation protocols were developed and implemented at all sites.

ELIGIBILITY:
Inclusion Criteria:

1. Individual with a genomic aberration identified by CMA, karyotyping, Southern blot analysis, PCR, FISH, and/or NGS or other standard of care (SOC) genetic testing technology whose clinical test results are available to compare with results from OGM.
2. Patients with prior negative SOC genetic testing results whose results are available to compare with results from OGM.

Exclusion Criteria:

1. Any individual who opted-out of research at the testing laboratory.
2. An individual whose genetic test contains the following variants: pathogenic sequence variants, abnormalities involving acrocentric p-arms and centromeres, below 20% for mosaicism, and tetraploidy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals will be recruited if they have standard of care genetic test results (such as CMA, karyotyping, Southern blot analysis, PCR, FISH, and/or NGS, etc.) to compare to optical genome mapping results.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity/Concordance and specificity of OGM with standard of care testing for detection of structural variants. | Through study completion, an average of 1 year
  OGM results are evaluated against the standard of care test and concordance (sensitivity and specificity) will be determined.

SECONDARY OUTCOMES:
Reproducibility and identification of structural variants beyond the limit of detection of standard of care methods. | Through study completion, an average of 1 year
  Inter-site as well as inter and intra-run variability of OGM will be assessed by reproducibility studies.

CONTACTS AND LOCATIONS:
Overall Officials: Alka Chaubey, PhD, FACMG, Principal Investigator — Bionano Genomics
Locations (8):
- United States (8):
  - Praxis Genomics, Atlanta, Georgia
  - Augusta University Research Institute, Augusta, Georgia
  - University of Iowa Hospitals & Clinics, Molecular Pathology, Iowa City, Iowa
  - Columbia University Irving Medical Center, New York, New York
  - DNA Microarray CGH Laboratory, Department of Pathology, University of Rochester Medical Center, West Henrietta, New York
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Lineagen (A Bionano Genomics Company), Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shieh JT, Penon-Portmann M, Wong KHY, Levy-Sakin M, Verghese M, Slavotinek A, Gallagher RC, Mendelsohn BA, Tenney J, Beleford D, Perry H, Chow SK, Sharo AG, Brenner SE, Qi Z, Yu J, Klein OD, Martin D, Kwok PY, Boffelli D. Application of full-genome analysis to diagnose rare monogenic disorders. NPJ Genom Med. 2021 Sep 23;6(1):77. doi: 10.1038/s41525-021-00241-5. PMID 34556655
- [Background] Stence AA, Thomason JG, Pruessner JA, Sompallae RR, Snow AN, Ma D, Moore SA, Bossler AD. Validation of Optical Genome Mapping for the Molecular Diagnosis of Facioscapulohumeral Muscular Dystrophy. J Mol Diagn. 2021 Nov;23(11):1506-1514. doi: 10.1016/j.jmoldx.2021.07.021. Epub 2021 Aug 9. PMID 34384893
- [Background] Mantere T, Neveling K, Pebrel-Richard C, Benoist M, van der Zande G, Kater-Baats E, Baatout I, van Beek R, Yammine T, Oorsprong M, Hsoumi F, Olde-Weghuis D, Majdali W, Vermeulen S, Pauper M, Lebbar A, Stevens-Kroef M, Sanlaville D, Dupont JM, Smeets D, Hoischen A, Schluth-Bolard C, El Khattabi L. Optical genome mapping enables constitutional chromosomal aberration detection. Am J Hum Genet. 2021 Aug 5;108(8):1409-1422. doi: 10.1016/j.ajhg.2021.05.012. Epub 2021 Jul 7. PMID 34237280
- [Background] Chaisson MJP, Sanders AD, Zhao X, Malhotra A, Porubsky D, Rausch T, Gardner EJ, Rodriguez OL, Guo L, Collins RL, Fan X, Wen J, Handsaker RE, Fairley S, Kronenberg ZN, Kong X, Hormozdiari F, Lee D, Wenger AM, Hastie AR, Antaki D, Anantharaman T, Audano PA, Brand H, Cantsilieris S, Cao H, Cerveira E, Chen C, Chen X, Chin CS, Chong Z, Chuang NT, Lambert CC, Church DM, Clarke L, Farrell A, Flores J, Galeev T, Gorkin DU, Gujral M, Guryev V, Heaton WH, Korlach J, Kumar S, Kwon JY, Lam ET, Lee JE, Lee J, Lee WP, Lee SP, Li S, Marks P, Viaud-Martinez K, Meiers S, Munson KM, Navarro FCP, Nelson BJ, Nodzak C, Noor A, Kyriazopoulou-Panagiotopoulou S, Pang AWC, Qiu Y, Rosanio G, Ryan M, Stutz A, Spierings DCJ, Ward A, Welch AE, Xiao M, Xu W, Zhang C, Zhu Q, Zheng-Bradley X, Lowy E, Yakneen S, McCarroll S, Jun G, Ding L, Koh CL, Ren B, Flicek P, Chen K, Gerstein MB, Kwok PY, Lansdorp PM, Marth GT, Sebat J, Shi X, Bashir A, Ye K, Devine SE, Talkowski ME, Mills RE, Marschall T, Korbel JO, Eichler EE, Lee C. Multi-platform discovery of haplotype-resolved structural variation in human genomes. Nat Commun. 2019 Apr 16;10(1):1784. doi: 10.1038/s41467-018-08148-z. PMID 30992455
- [Background] Chan S, Lam E, Saghbini M, Bocklandt S, Hastie A, Cao H, Holmlin E, Borodkin M. Structural Variation Detection and Analysis Using Bionano Optical Mapping. Methods Mol Biol. 2018;1833:193-203. doi: 10.1007/978-1-4939-8666-8_16. PMID 30039375
- [Background] Barseghyan H, Tang W, Wang RT, Almalvez M, Segura E, Bramble MS, Lipson A, Douine ED, Lee H, Delot EC, Nelson SF, Vilain E. Next-generation mapping: a novel approach for detection of pathogenic structural variants with a potential utility in clinical diagnosis. Genome Med. 2017 Oct 25;9(1):90. doi: 10.1186/s13073-017-0479-0. PMID 29070057
- [Background] Lam ET, Hastie A, Lin C, Ehrlich D, Das SK, Austin MD, Deshpande P, Cao H, Nagarajan N, Xiao M, Kwok PY. Genome mapping on nanochannel arrays for structural variation analysis and sequence assembly. Nat Biotechnol. 2012 Aug;30(8):771-6. doi: 10.1038/nbt.2303. PMID 22797562
- [Result] Iqbal MA, Broeckel U, Levy B, Sinner S, Sahajpal N, Rodriguez V, Stence A, Awayda K, Scharer G, Skinner C, Stevenson R, Bossler A, Nagy PL, Kohle R. Multi-site technical performance and concordance of optical genome mapping: constitutional postnatal study for SV, CNV, and repeat array analysis. MedRxiv (pre-print). 2021 Dec 30; doi: https://doi.org/10.1101/2021.12.27.21268432